CLINICAL TRIAL: NCT01985113
Title: Correlation Study of Blood and Tissue Thioredoxin Reductase Activity in Early Stage On-small Cell Lung Cancers
Brief Title: Correlation Research of Thioredoxin Reductase in Lung Cancer
Acronym: TRCRLC
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Nong Yang, chief, Hunan Province Tumor Hospital
Other Study IDs: TR001; TRRFLC1 (Other: HunanPTH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-small Cell Lung Cancer; Benign Neoplasm of Lung
Keywords: thioredoxin reductase; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue and lung benign mass are obtained in surgery, and blood serum before surgery and 3-5 days after surgery, blood should be taken and centrifuged then stored at -20 degree, tumor tissue and lung benign mass should be stored at -180 degree within 5 mins during surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- early staged non-small cell lung cancers: patients who diagnosed as early staged non-small cell lung cancer after surgery
- lung benign mass patients: patients who diagnosed as lung benign mass after surgery

SUMMARY:
In pre-clinical study the investigators found that the thioredoxin reductase activity of serum harbours huge difference between cancer patients and non-cancer patients, the enzyme activity elevated remarkably among cancer patients, so the investigators hypothesis that this is due to tumor cells loading of the patients, the enzyme activity may harbours huge difference between carcinoma tissues and para-carcinoma tissues in early staged non-small cell lung cancers, and after surgery, the enzyme activity may fall down to a normal level because of removing of tumor.

DETAILED DESCRIPTION:
This is a cooperative research project in Thoracic Surgery Department and Medical Oncology Department of Affiliated Cancer Hospital of xiangya School of Medicine Central South University, and the State Key Laboratory for Natural Medicine and Biomimetic Drugs Perking University. The primary objective is to measure the thioredoxin reductase activity using blood and lung cancer tissue and measure thioredoxin reductase messenger ribonucleic acid (mRNA) and protein expression using lung cancer and pericarcinomatous tissue in early staged(Ⅰ~ⅢA) non-small lung cancers, to study the correlations of thioredoxin reductase between blood and tissue. The secondary objectives are to measure the thioredoxin reductase activity between non small lung cancers and lung benign lesion patients to identify the difference between tumor and lung benign mass.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven staged(Ⅰ~ⅢA) non-small cell lung cancer or CT scan shows resectable lung mass
* Receive surgery in Thoracic Oncology department Hunan Tumor Hospital without contraindication of surgery
* Malignant tumor treatment naive（except for surgery for cervical cancer and cutaneous squamous cell carcinoma 5 years before）
* Signed informed consent about providing blood and tissue for study

Exclusion Criteria:

* Patients have received antitumor treatment
* Patients with contraindication of surgery or patients who need adjuvant chemotherapy with contraindication of chemotherapy
* Pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early staged NSCLC and lung benign lesion Patients show resectable lung mass in CT scan, suspected lung cancer and receive surgery in Affiliated Cancer Hospital of Xiangya School of Medicine Central South University
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2013-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
measure the thioredoxin reductase activity in blood, tumor and pericarcinomatous tissue | blood should be taken in 2 days before surgery, tumor and pericarcinomatous tissues should be stored and tested in one month
  3-4 ml blood should be taken and centrifuged in 30 mins, then the serum should be stored at -20 degree, then serum thioredoxin reductase activity should be measured in one month. Tumor and pericarcinomatous tissues should be stored at -180 degree and enzyme activity should be measured within one month

SECONDARY OUTCOMES:
Measure the difference of thioredoxin reductase activity between lung cancer tissue and lung benign mass | Tumor tissue or lung benign mass obtained during surgery should be stored at -180 degree within 5 mins and enzyme activity should be measured within one month
  Tumor tissue or lung benign mass obtained during surgery should be stored at -180 degree within 5 mins and enzyme activity should be measured within one month.
Measure the thioredoxin reductase mRNA and protein expression in tumor and pericarcimomatous tissue | Tumor tissue or pericarcimomatous tissue should be stored at -180 degree, then qRT-PCR should be done within 3 months
  Tumor tissue or pericarcimomatous tissue should be stored at -180 degree, then qRT-PCR should be done within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nong Yang, MD, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China